CLINICAL TRIAL: NCT00724750
Title: Prospective Randomized Control Trial Comparing Two Methods of Negative Pressure Wound Therapy: Gauze Suction Versus Vacuum Assisted Closure Device
Brief Title: Comparison of Two Methods of Negative Pressure Wound Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14817A
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Acute Wounds From Trauma; Dehiscence or Surgical Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-SUC (Experimental): Gauze suction (G-SUC) Negative Pressure Wound Therapy, continuous wall suction at 75 to 80 mm Hg was applied and dressings were changed daily.
  Interventions: Device: Gauze suction (G-SUC)
- Vacuum Assisted Closure (Active Comparator): Vacuum Assisted Closure Device (VAC) Negative Pressure Wound Therapy, continuous suction at 75 to 125 mm Hg and the dressing was changed every 48 hours.
  Interventions: Device: Vacuum Assisted Closure Device (VAC)

INTERVENTIONS:
Device: Gauze suction (G-SUC) — Negative pressure wound therapy
  Arms: G-SUC
Device: Vacuum Assisted Closure Device (VAC) — Negative Pressure Wound Therapy
  Arms: Vacuum Assisted Closure

SUMMARY:
The current standard for negative pressure wound therapy is the Vacuum Assisted Closure Device (VAC), a commercial system that utilizes a computerized suction pump to apply negative pressure to an open-cell poly-urethane foam dressing sealed over a wound. The VAC system is effective but has some drawbacks:

* The system is expensive.
* There us conflicting data about the effectiveness of VAC therapy for infected wounds.
* VAC therapy is difficult to use (and frequently fails) in wounds with excess fluid drainage, and in wounds near body orifices.

Over the past 4 years, we have accumulated additional experience with negative pressure wound therapy using wall suction applied to sealed gauze dressings with about 30 patients. We call this method G-SUC and have used it when we have been unable to maintain a dressing seal with the VAC system (due to excess drainage or wound location), for management if infected wounds. We have found this method to be effective without any specific negative side effects.

Our specific aims are:

1. Compare the effectiveness of G-SUC and standard VAC therapy. Outcomes measured for each method will include the proportional change in wound size over 1 - 2 weeks.
2. Compare the effectiveness of G-SUC and VAC system in controlling wound infections as measured by the number of patients who are able to clear infection by 4 days.
3. Compare the failure of each method of therapy by documenting the number of dressing that cannot be maintained because of fluid or suction.
4. Measure and compare the cost of wound treatment with the two methods including direct cost and time spent at the bed side performing the dressing change.

Our hypotheses are:

1. G-SUC and VAC are equivalent for the treatment of uncomplicated wounds in the acute care, in-patient setting.
2. G-SUC is more effective than VAC for management of infected wounds.
3. G-SUC is more versatile than VAC, and functional G-SUC dressings can be maintained in situations where functional VAC dressings cannot.
4. Negative pressure therapy with G-SUC is less costly than VAC.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized patients at the University of Chicago Medical Center with acute wounds resulting from ether trauma, dehiscence or surgical complications

Exclusion Criteria:

* Patients with systemic sepsis caused by wound infection
* Those with grossly necrotic wounds
* Malignancy in the wound
* Wounds with untreated osteomyelitis
* Patients with allergy to sulfamylon and Dakin's (sodium hypochlorite) Patients with 2 first criteria would become eligible once their sepsis resolves and/or necrotic tissue has been debrided from the wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Gottlieb, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Dorafshar AH, Franczyk M, Gottlieb LJ, Wroblewski KE, Lohman RF. A prospective randomized trial comparing subatmospheric wound therapy with a sealed gauze dressing and the standard vacuum-assisted closure device. Ann Plast Surg. 2012 Jul;69(1):79-84. doi: 10.1097/SAP.0b013e318221286c. PMID 21712704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | G-SUC | Vacuum Assisted Closure
Started | 45 | 42
Completed | 45 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-SUC | Vacuum Assisted Closure | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Continuous [Mean (Full Range); unit: years] | 53 [23 to 80] | 54 [19 to 82] | 53 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 14 | 19 | 33
Region of Enrollment [Number; unit: participants]
  United States | 45 | 42 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percent Change Per Day in Wound Surface Area
Description: Wound surface area was measured daily. The percent change from Day 1 was calculated. A negative value indicates a decrease.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: % change per day
Arm/Group | G-SUC | Vacuum Assisted Closure
Number analyzed (Participants) | 45 | 42
% change per day | -4.5 [-5.3 to -3.8] | -4.9 [-6.0 to -3.8]
Statistical Analysis 1: Comparison: G-SUC vs Vacuum Assisted Closure; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 5%/day. For 80% power and a significance (alpha) level of 0.05; and assuming a common standard deviation of 9%, 41 subjects per group were needed; p = 0.60, Mixed Models Analysis — The rate of change for the 2 groups was compared by testing the treatment-by-time interaction in the model

2. Primary Outcome: Percent Change Per Day in Wound Volume
Description: Wound volume was measured daily. The percent change from Day 1 was calculated. A negative value indicates a decrease.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: % change per day
Arm/Group | G-SUC | Vacuum Assisted Closure
Number analyzed (Participants) | 45 | 42
% change per day | -8.4 [-9.5 to -7.2] | -9.8 [-11.5 to -8.1]
Statistical Analysis 1: Comparison: G-SUC vs Vacuum Assisted Closure; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 5%/day; p = 0.19, Mixed Models Analysis — The rate of change for the 2 groups was compared by testing the treatment-by-time interaction

3. Secondary Outcome: Failure to Maintain Dressing Because of Fluid or Suction Leaks
Time Frame: Participants were followed for the duration of inpatient stay, an average of 5 days.
Measure: Number; unit: participants
Arm/Group | G-SUC | Vacuum Assisted Closure
Number analyzed (Participants) | 45 | 42
participants | 0 | 4

4. Secondary Outcome: Average Time Spent on Dressing Changes
Description: Time was measured from the start of the dressing change until the initiation of suction.
Time Frame: Participants were followed for the duration of inpatient stay, an average of 5 days.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-SUC | Vacuum Assisted Closure
Number analyzed (Participants) | 45 | 42
minutes | 19 (6) | 31 (13)
Statistical Analysis 1: Comparison: G-SUC vs Vacuum Assisted Closure; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Pain Score With Dressing Changes
Description: Self-reported pain levels were used to assess pain. Patients were asked to rate their pain level according to the 0 to 10 linear analog scale immediately before, during, and after removal of the dressing. The average number of dressing changes for the G-SUC group was 4.5 (range 2-15) and the average number of dressing changes for the VAC group was 2.8 (range 2-6). The sum of pain intensity differences (SPID) was used to facilitate comparison of pain levels. The SPID score was calculated for each dressing change using the formula: (pain during - pain before) + (pain after - pain during). Higher values indicating greater pain.
Time Frame: Participants were followed for the duration of inpatient stay, an average of 5 days.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | G-SUC | Vacuum Assisted Closure
Number analyzed (Participants) | 45 | 42
units on a scale | 0.50 [-0.11 to 1.11] | 1.73 [0.91 to 2.54]
Statistical Analysis 1: Comparison: G-SUC vs Vacuum Assisted Closure; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

6. Secondary Outcome: Average Cost of Supplies and Rental
Description: Direct costs for each type of dressing were measured. In the VAC group, this included rental charges for the equipment and the cost of supplies. In the G-SUC group, this included the cost of supplies (suction canisters, catheters or drains, tubing, gauze, and adhesive drapes).
Time Frame: Participants were followed for the duration of inpatient stay, an average of 5 days.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | G-SUC | Vacuum Assisted Closure
Number analyzed (Participants) | 45 | 42
dollars | 4.22 (1.57) | 96.51 (11.26)
Statistical Analysis 1: Comparison: G-SUC vs Vacuum Assisted Closure; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | G-SUC | Vacuum Assisted Closure
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/42
Other Adverse Events (participants affected / at risk) | 0/45 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-SUC (N=45) | Vacuum Assisted Closure (N=42)
Hematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes